CLINICAL TRIAL: NCT04009850
Title: Impact of Cigarette and E-cigarette Flavors on Adult Smoking Behavior
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study enrollment was temporarily paused in 2020 due to COVID-19. Study was closed without further enrollment in 2022.
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000025572; 2U54DA036151-06 (NIH)
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: Within-subject design comparing smoking behavior when using menthol vs. non-menthol cigarettes with either menthol or tobacco flavored e-cigarettes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menthol e-cigarette (Experimental): Adult smokers will be switched from using menthol cigarettes to non-menthol cigarettes and a menthol flavored e-cigarette
  Interventions: Other: Cigarette Brand Switching
- Tobacco e-cigarette (Experimental): Adult smokers will be switched from using menthol cigarettes to non-menthol cigarettes and a tobacco flavored e-cigarette
  Interventions: Other: E-cigarette Flavor

INTERVENTIONS:
Other: Cigarette Brand Switching — Adult smokers will be switched from smoking menthol cigarettes to non-menthol cigarettes
  Arms: Menthol e-cigarette
Other: E-cigarette Flavor — Adult smokers will be provided with either menthol or tobacco flavored e-cigarettes in addition to the non-menthol cigarettes
  Arms: Tobacco e-cigarette

SUMMARY:
This study will investigate within-person changes in smoking behavior when current menthol smokers are switched to non-menthol cigarettes and either tobacco or menthol flavored e-cigarettes.

DETAILED DESCRIPTION:
The goals of this project include evaluating within-subject changes in cigarette satisfaction and smoking behavior after switching from menthol cigarettes and investigating whether outcomes differ between subjects based on use of menthol vs. tobacco flavored e-cigarettes. Within-person changes in cigarette satisfaction and smoking behavior will be assessed during the last week of the non-menthol cigarette smoking period compared to the menthol cigarette smoking period. Preference and use of both the cigarette and e-cigarette products during the switching period will be compared and the extent to which menthol flavored (vs. tobacco) e-cigarettes are preferred among menthol smokers will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Able to read English
* Cigarette smoker

Exclusion Criteria:

* Seeking smoking cessation treatment
* Serious psychiatric or medical condition
* Use of other drugs
* Unable or unwilling to complete study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-09 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krysten Bold, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Menthol E-cigarette | Tobacco E-cigarette
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in the tobacco e-cigarette condition prior to study termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Menthol E-cigarette | Tobacco E-cigarette | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (13.6) |  | 43.3 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 2 |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 3 |  | 3
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 2 |  | 2
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Cigarettes Smoked
Description: Self-reported total number of cigarettes smoked per day (Timeline Follow Back)
Time Frame: Week 6
Population: No participants were enrolled in the tobacco e-cigarette condition.
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Menthol E-cigarette | Tobacco E-cigarette
Number analyzed (Participants) | 3 | 0
cigarettes per day | 19 (16) |

2. Secondary Outcome: E-cigarette Use
Description: Self-reported e-cigarette use compared by e-cigarette flavor (Timeline Follow Back)
Time Frame: Week 6
Population: Analyses were not conducted for this outcome examining use by e-cigarette flavor condition because no participants were enrolled in the tobacco e-cigarette condition.
Arm/Group | Menthol E-cigarette | Tobacco E-cigarette
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Tobacco Product Satisfaction
Description: Self-reported subjective ratings of satisfaction with tobacco products (Modified Cigarette/E-cigarette Evaluation Questionnaire), rated 1-7 with higher scores indicating greater satisfaction
Time Frame: Week 6
Population: No participants were enrolled in the tobacco e-cigarette condition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Menthol E-cigarette | Tobacco E-cigarette
Number analyzed (Participants) | 3 | 0
units on a scale | 1.7 (1.6) |

4. Secondary Outcome: Motivation to Quit Smoking
Description: Self-reported motivation to quit smoking cigarettes (Contemplation Ladder), rated 1-10, higher scores indicate greater motivation to quit
Time Frame: Week 6
Population: No participants were enrolled in the tobacco e-cigarette condition.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Menthol E-cigarette | Tobacco E-cigarette
Number analyzed (Participants) | 3 | 0
units on a scale | 7.7 (2.1) |

5. Secondary Outcome: Nicotine Dependence
Description: Self-reported nicotine dependence (NIH Promis Dependence Measure), rated 1-5, higher scores indicate greater dependence
Time Frame: Week 6
Population: No participants were enrolled in the tobacco e-cigarette condition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Menthol E-cigarette | Tobacco E-cigarette
Number analyzed (Participants) | 3 | 0
score on a scale | 3.8 (1.1) |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the 10 weeks of study participation.
Description: No participants were enrolled in the tobacco e-cigarette condition.
Arm/Group | Menthol E-cigarette | Tobacco E-cigarette
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT04009850/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT04009850/ICF_001.pdf